CLINICAL TRIAL: NCT07281248
Title: TRIMODAL PREHABILITATION PROGRAM IN PATIENTS WITH GASTROINTESTINAL CANCER DURING NEOADJUVANT TREATMENT: A PILOT STUDY
Brief Title: TRIMODAL PREHABILITATION IN GASTROINTESTINAL CANCER
Acronym: PREDIGEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Ana Ruiz-Casado, PRINCIPAL INVESTIGATOR, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PREH-PHM-03; SEOM (Other Grant/Funding Number: SEOM)
Record Dates: First submitted 2025-08-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Digestive Neoplasms
Keywords: cancer; prehabilitation; gastrointestinal; exercise; trimodal
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: All the participants will receive trimodal prehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): Gastrointestinal cancer patients will participate in a trimodal prehabilitation program, including nutrition, psychological support, and exercise interventions.
  Interventions: Combination Product: TRIMODAL PREHABILITATION

INTERVENTIONS:
Combination Product: TRIMODAL PREHABILITATION — Gastrointestinal cancer patients (not stage 4) will undergo trimodal prehabilitation: nutrition, psychological, and exercise support.

SUMMARY:
Digestive cancers account for a substantial proportion of oncological patients, representing over 20% of cases treated in hospitals, and are generally managed through a multidisciplinary approach that has markedly improved survival outcomes over recent decades. Surgical resection remains the cornerstone of curative treatment, often preceded by neoadjuvant chemotherapy, radiotherapy, or combined modalities. Notably, a significant proportion of patients eligible for abdominal surgery are older adults, with approximately one in three being over 75 years of age. Advances such as Enhanced Recovery After Surgery (ERAS) protocols and the centralization of complex surgical procedures have contributed to better outcomes, including higher rates of radical resections, improved survival, reduced postoperative complications, and shorter hospital stays.

While some risk factors are non-modifiable, such as age, sex, tumor stage, comorbidities, and tumor biology, several modifiable factors can be optimized prior to surgery to improve postoperative outcomes. These include smoking cessation, enhancement of aerobic capacity and muscular strength, nutritional optimization, emotional resilience, and correction of anemia or other metabolic derangements. Preoperative exercise, ideally embedded within a multimodal prehabilitation program, is recommended for all patients undergoing major surgery. The neoadjuvant period represents a valuable window to implement trimodal prehabilitation strategies encompassing physical exercise, nutritional support, and psychological interventions, aimed at reducing postoperative complications, shortening hospital length of stay, and improving functional recovery.

Physical fitness in this context is multidimensional, encompassing aerobic capacity, muscle strength, and body composition. Aerobic capacity predicts postoperative complications and length of hospital stay, while low muscle strength and sarcopenia are associated with higher morbidity and poorer prognosis. Inspiratory muscle training can further reduce pulmonary complications and accelerate recovery. Nutritional status is a critical determinant of surgical outcomes in gastrointestinal cancer, with malnutrition affecting up to 80% of patients at diagnosis. Comprehensive assessment, including dietary intake, anthropometric measurements, physical examination, and biomarkers such as albumin and transferrin, is essential, and targeted interventions including protein supplementation, pancreatic enzyme replacement, or tailored dietary strategies should be implemented when indicated. Body composition, particularly sarcopenia and cachexia, is closely linked to both nutrition and exercise, and can be assessed through imaging techniques such as DXA, CT, or MRI, or via bioelectrical impedance in research settings, with simpler bedside assessments used in clinical practice.

Emotional wellbeing also plays a significant role, as preoperative anxiety and depression can negatively influence recovery, adherence to rehabilitation, and overall quality of life. Psychological support, stress management, and behavioral interventions can improve patient engagement and enhance outcomes. The physiological principles of hormesis and cross-stressor adaptation suggest that controlled exercise can improve resilience to both physical and psychological stressors, including the stress of surgery itself. Additional modifiable factors such as absolute cessation of alcohol and tobacco, glycemic control in diabetic patients, correction of anemia (including iron deficiency), and frailty assessment in older adults are critical components of preoperative optimization.

Major abdominal surgery carries substantial risk, including infections, bleeding, and anastomotic complications, which directly impact quality of life and lengthen hospitalization. Evidence from randomized controlled trials indicates that multimodal prehabilitation effectively reduces postoperative complications and shortens hospital stay. However, motivating patients to engage in exercise during neoadjuvant therapy can be challenging due to treatment-related fatigue, nausea, and other side effects. Integrating behavioral theories such as Self-Determination Theory and the Theory of Planned Behavior can enhance intrinsic motivation by fostering autonomy, competence, and relatedness, and addressing attitudes, subjective norms, and perceived behavioral control, ultimately promoting adherence to prehabilitation programs and optimizing postoperative recovery.

DETAILED DESCRIPTION:
9. INTERVENTION PHYSICAL PREHABILITATION PROGRAMME Prior to the intervention, a complete physical assessment will be carried out. In addition, a motivational interview will be conducted, which is a promising technique for addressing many types of behavioural changes in cancer patients or survivors.

The training will consist of two main components (cardiorespiratory endurance and muscle strength) and two secondary components (flexibility and balance). A plan will be followed to increase the intensity of the training in relation to the patients' tolerance and functional capacity.

AEROBIC EXERCISE: A frequency of at least 5 days per week should be achieved in the case of moderate exercise and at least 2 days in the case of vigorous exercise, aiming for a total of 150-300 minutes of moderate-vigorous physical activity or 75-150 minutes in the case of vigorous activity (WHO, 2020). Moderate intensity is considered to be training at 40-59% of peak oxygen consumption reserve (the difference between consumption at maximum exercise and at rest), or training at 55-69% of maximum HR or 6-7 on the Borg scale. Vigorous intensity is considered to be training at 60-84% of peak oxygen consumption, or training at 70-89% of maximum HR or 8-9 on the Borg scale.

The type of aerobic exercise will differ depending on the stage of the patient's treatment and their tolerance. When exercising independently, they can do most of the exercise by walking and cycling (which trains the large muscle groups). If their physical condition allows it, they could do interval training. If the patient tolerates it, the intensity can be increased, but it must be remembered that as they progress in training, they also progress in chemotherapy treatment and their tolerance to exercise decreases.

In the supervised part, the training methodology will be varied (i.e. circuits with different activities, games, etc.) in order to avoid monotony and boredom, which have been linked to lower motivation to engage in physical activity. In any case, training will be planned and periodised on a day-to-day basis in order to adapt the training sessions to the individual needs of each patient.

STRENGTH TRAINING: Two supervised sessions per week should be carried out, which will include an individualised progression from single-joint exercises to multi-joint exercises. Initially, priority will be given to the volume and subsequently to the intensity of the training. There will be a daily schedule based on the patient's daily capacity due to the effect of the treatment and their physical condition. Therefore, different adaptations will be designed, and the patient will be able to choose the training that best suits that day, all of which will meet the training objectives included in the prehabilitation programme. With a Borg scale rating of 7-8. Flexibility and balance exercises will be recommended.

INSPIRATORY MUSCLE TRAINING: 5 weekly sessions of 15 minutes, with an initial load of 20-30% of maximum inspiratory pressure until reaching 60%. The first sessions will always be supervised. Expiratory muscles-vagus nerve: Patients will be taught to breathe at a slow pace for 5 minutes. Breathing will be performed using biased patterns: Inhale and count 1-5. Hold your breath and count 1-2. Exhale and count 1-7.

In our first programme, we were able to demonstrate that supervised exercise during very demanding chemotherapy treatment such as FOLFIRINOX was feasible and achieved very high adherence and a very good recruitment rate. For this reason, in this programme we have increased the adherence requirements to consider it feasible. 100% adherence will be adherence to all sessions.

The face-to-face training sessions will take place on Tuesdays and Thursdays at the 'Terra' cross-fit space in Majadahonda.

NUTRITIONAL PREHABILITATION PROGRAMME The nutrition specialist must understand each subject's diet and identify any nutritional deficiencies that may be occurring. They must help the patient to optimise their nutrition. It is critical to identify malnourished patients, in which case nutritional supplements will be provided by the responsible physicians. Nutritional support will be in line with international recommendations. Follow-up by a nutrition specialist will be guaranteed with monthly sessions, which may be increased if a high risk of nutritional compromise is identified.

The consumption of protein after strength training sessions should be promoted within the prehabilitation programme.

PSYCHOLOGICAL PREHABILITATION PROGRAMME The psychologist will identify those patients who require psychological intervention. The aim of the psychologist's intervention is twofold. On the one hand, they will try to achieve high adherence to the prehabilitation programme and, on the other, they will prepare the patient to face complex surgery. Psychological support will be guaranteed during prehabilitation in monthly sessions, which may be conducted individually or in groups.

EXTRACTION OF BIOLOGICAL SAMPLES Blood samples will be taken at baseline and before surgery to study aspects related to the programme in the future, depending on findings and future funding.

In addition, the possibility of taking blood samples before and after the first training session will be explored

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* ECOG 0-2
* Being able to complete the mile-time test
* Stages I-III
* Being able to understand the informed consent
* Gastrointestinal cancer diagnosed

Exclusion Criteria:

* Metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the feasibility of a trimodal prehabilitation program with motivational strategies during chemotherapy in a multidisciplinary hospital setting. | 1 year
  Feasibility will be assessed based on the rejection rate (<50%) and adherence (>50%). Adherence will be considered according to the training options. There are two sessions per week (attendance at four sessions in a 15-day cycle, 100%, etc.).

SECONDARY OUTCOMES:
Changes in (estimated) cardiorespiratory fitness | 3-6 months (from 1st treatment to surgery)
  One-mile walking test (in meters). (Rockport test) A higher distance means a worse result.
Changes in muscle strength | 3-6 months (from 1st treatment to surgery)
  Handgrip dynamometer test
Changes in body composition | 3-6 months (from 1st treatment to surgery)
  body mass index
Changes in levels of physical activity at week | 3-6 months (from 1st treatment to surgery)
  By accelerometers (counts)
Changes in quality of life | 3-6 months (from 1st treatment to surgery)
  Global quality of life questionnaire (EORTC-QLQ30)
Changes in fatigue levels | 3-6 months (from 1st treatment to surgery)
  The PERFORM questionnaire (PQ) (12-60). A higher score means a lower fatigue level.
Dose intensity in neoadjuvant treatment | three months
  percentage of intended doses that are administered in the due time
Describe post-surgical complications | 3-6 months (from 1st treatment to surgery)
  Surgical wound and pancreatic fistula. Postoperative complications according to Clavien-Dindo (CCI score). Comprehensive Complication Index CCI SCORE: summarizes postoperative well-being concerning complications according to the Clavien Dindo classification.
Describe psychological status | 3-6 months (from 1st treatment to surgery)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire used to screen for psychological distress, specifically anxiety and depression, in adult patients. It consists of two subscales-one for anxiety (HADS-A) and one for depression (HADS-D)-with each of the 14 items rated on a four-point scale from 0 to 3, resulting in a maximum score of 21 for each subscale.
To describe body composition | 3-6 months (from 1st treatment to surgery)
  Weight and height will be measured to define body mass index (kg/m2)
Percentage of pathological complete responses | 4-6 weeks after surgery
  Percentage of patients with no viable cells in the surgical specimen
Hindrances and facilitators of patients | 3-6 months (from 1st treatment to surgery)
  Qualitative methods will be used to complete the information provided by quantitative methods. After the exercise program, each patient will be interviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ruiz Casado Principal Investigator, PhD, MD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Madrid, Spain